CLINICAL TRIAL: NCT04403074
Title: Endoscopic Ultrasound-Guided Celiac Plexus Neurolysis (EUS-CPN) for Chronic Pancreatitis, Database Repository
Brief Title: Endoscopic Ultrasound-Guided Celiac Plexus Neurolysis (EUS-CPN) for Chronic Pancreatitis
Acronym: CPN
Status: Recruiting | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Mohammad Al-Haddad, Associate Professor of Medicine, Associate Clinical Director, Indiana University
Other Study IDs: 1708591420
Record Dates: First submitted 2018-10-10; First posted 2020-05-27 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Chronic Pancreatitis
Keywords: Pancreatitis; Indiana; Block; Celiac; Plexus
MeSH Terms: conditions — Pancreatitis, Chronic; Pancreatitis; Bites and Stings; Celiac Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic Pancreatitis Patients: Patients that have Chronic Pancreatitis and the current treatment with Celiac Plexus Blocks (CPB) are providing minimal relief of pain (CPB provide less than one month of pain relief). These patient will then receive a Celiac Plexus Neurolysis.
  Interventions: Procedure: Celiac Plexus Neurolysis

INTERVENTIONS:
Procedure: Celiac Plexus Neurolysis — When CPBs are not effective (less than one month of relief) then a Celiac Plexus Neurolysis may be completed to manage pain associated with Chronic Pancreatitis.

SUMMARY:
Physicians need a tracking system for specific treatment modalities, and data to determine the impact of endoscopic ultrasound pain management for patients with chronic pancreatitis.

DETAILED DESCRIPTION:
Chronic pancreatitis is extremely painful and pain management in patients with chronic pancreatitis is challenging. The etiology of abdominal pain in chronic pancreatitis is considered multifactorial. Current treatments for pain control primarily include narcotic & opioid administration; however, these medications require titration of dosage for optimal pain control and are frequently followed by adverse effects such as constipation, nausea or drug addiction. Currently, the FDA has imposed strict regulations regarding the amount, frequency & length of time patients may receive these medications. With tightly controlled regulations for prescribing narcotics and opioids for chronic pain management, the epidemic of street drug usage and overdose has dramatically increased. Alternatively, celiac plexus block and celiac plexus neurolysis performed under EUS guidance have been employed for pain control for at least 2 decades and deemed safe. Celiac plexus block refers to temporary inhibition of nerves of the celiac plexus, by using a combination of steroid and numbing medications injected into the celiac plexus ganglia. Celiac plexus neurolysis (CPN) refers to a temporary to semi-permanent inhibition of nerves of the celiac plexus ganglia. Injection of alcohol as a neurolytic agent is used in place of the steroid which causes neurolysis of the celiac plexus or ganglia.

This study will focus on collecting data related to endoscopic ultrasound procedures performed by Indiana University EUS physicians; specifically for the management of chronic pancreatitis pain. This data will be used for research purposes to determine the clinical impact of EUS-CPN management in chronic pancreatitis pain. The physicians will also be able to better understand the patient's condition and disease process that may lead to improved patient management.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Referral for the treatment of pain related to chronic pancreatitis

Exclusion Criteria:

* Less than 18 years of age
* Absence of chronic pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: As long as patients fall under the inclusion criteria and do not fall under exclusions, every patient can be considered. Patient must be declared safe to undergo procedure on individual basis from an evaluation from head doctor on study.
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2017-10-20 (Actual); Primary Completion 2029-10-20 (Estimated); Study Completion 2029-10-20 (Estimated)

PRIMARY OUTCOMES:
Use of Pain medication | Immediately post procedure & weekly up to 24 weeks
  Use of pain medication (by using morphine equivalents) for each patient will be tracked weekly for up to 24 weeks post CPN to track pain management/relief for the of patients. There should be a lessening in use of pain medication as time progesses.
Patient's pain intensity score (numeric pain rating scale using the visual analogue scale VAS from 1-10) will be assessed weekly (via phone call follow ups) starting right after CPN and continuing for 24 weeks. | Immediately post procedure and weekly up to 24 weeks
  Compare weekly pain intensity score for pain management/relief of patients.
Dosage of pain medication | Immediately post procedure and weekly up to 24 weeks
  Compare dose of pain medication post procedure & weekly for up to 24 weeks after converting all to morphine equivalents

CONTACTS AND LOCATIONS:
Overall Officials: Mo A, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States